CLINICAL TRIAL: NCT03973151
Title: A Phase I/II, Single Arm, Dose Escalation and Cohort Expansion Study to Evaluate Safety, Preliminary Efficacy of HL-085 in Patients With NRAS Mutant Advanced Melanoma
Brief Title: Study of HL-085 in NRAS Mutant Advanced Melanoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Kechow Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HL-085-101
Record Dates: First submitted 2017-12-19; First posted 2019-06-04 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Melanoma
Keywords: Melanoma; NRAS
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HL-085 (Experimental): HL-085 will be administered as BID with specified dose.
  Interventions: Drug: HL-085

INTERVENTIONS:
Drug: HL-085 — HL-085 is one MEK inhibitor.

SUMMARY:
This is a phase I/II, open-label, dose escalation study to evaluate tolerability, safety, pharmacokinetics and efficacy in patients with NRAS mutant advanced melanoma .

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed unresectable Stage III or Stage IV melanoma according to AJCC (Version 7, 2010).
2. Subjects must have NRAS mutation in melanoma.
3. Chemotherapy, immunotherapy or radiotherapy ≥ 4 weeks prior to starting the study treatment. Surgery (except for tumor biopsy) or severe trauma ≤ 14 days prior to starting the study treatment.
4. ECOG performance status of 0-1.
5. Life expectancy ≥ 3 months.
6. Ability to take the medicine orally.
7. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Prior therapy with a MEK-inhibitor
2. Patients with known hypersensitivity to study drug ingredients or their analogues.
3. Active central nervous system (CNS) lesion.
4. ECG QTcB≥480msec in screening, or history of congenital long QT syndrome.
5. Subjects with bleeding symptoms at Grade 3 (NCI-CTCAE v4.03) within 4 weeks prior to starting study treatment.
6. Uncontrolled concomitant diseases or infectious diseases.
7. Retinal diseases (Retinal Vein Occlusion (RVO) or Retinal pigment epithelial detachment (RPED) , et al.).
8. History of HIV,HCV,HBV infection.
9. Interstitial lung disease or interstitial pneumonitis, including clinically significant radiation pneumonitis will be excluded.
10. Serum HCG test is positive.
11. Other conditions that influence the results and increase the risk of study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2021-01-18 (Actual); Study Completion 2021-01-18 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | Duration of the study, estimated to be approximately 24 months.
  Number of Treatment-Related Adverse Events as Assessed by CTCAE v4.03 during the study period
Maximum tolerated dose (MTD) | DLTs within the first cycle of therapy (up to 35 days)
  The dose level immediately below the dose level at which ≥ 2 patients from a cohort of 3 to 6 patients experience a dose-limiting toxicity (DLT)

SECONDARY OUTCOMES:
Objective Response Rate (ORR) as measure of efficacy | Duration of the study, estimated to be approximately 24 months.
  Efficacy estimated as the Objective Response Rate (ORR) , which is the sum of Partial Response (PR) and Complete Response (CR) as determined by RECIST 1.1
Area under the plasma concentration versus time curve (AUC) | Duration of the study, estimated to be approximately 24 months
  AUC of HL-085 following single and repeated dosing
Peak Plasma Concentration (Cmax) | Duration of the study, estimated to be approximately 24 months
  Cmax of HL-085 following single and repeated dosing
Time to maximum observed plasma drug concentration (Tmax) | Duration of the study, estimated to be approximately 24 months.
  Tmax of HL-085 following single and repeated dosing
Half-life (T1/2) | Duration of the study, estimated to be approximately 24 months.
  T1/2 of HL-085 following single and repeated dosing

CONTACTS AND LOCATIONS:
Overall Officials: Hongqi Tian, Ph.D, Study Director — Shanghai Kechow Pharma, Inc.
Locations (2):
- China (2):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wang X, Luo Z, Chen J, Chen Y, Ji D, Fan L, Chen L, Zhao Q, Hu P, Sun P, Jia Z, Guo J, Si L. First-in-human phase I dose-escalation and dose-expansion trial of the selective MEK inhibitor HL-085 in patients with advanced melanoma harboring NRAS mutations. BMC Med. 2023 Jan 4;21(1):2. doi: 10.1186/s12916-022-02669-7. PMID 36600247